CLINICAL TRIAL: NCT02883569
Title: Randomized Control Trial. Comparative Effectiveness Study for Surgery vs. Non-Surgery in Patients With Low Back Pain
Brief Title: Comparative Effectiveness Study for Surgery vs. Non-Surgery in Patients With Low Back Pain
Acronym: CES_SNS_LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Gangnam Severance Hospital (Other); Severance Hospital (Other); Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Chun Kee Chung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LBP
Record Dates: First submitted 2016-07-25; First posted 2016-08-30 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Low Back Pain
Keywords: Low back pain; Intervertebral Disc Degeneration; Spinal stenosis; Comparative Effectiveness Research; Cost-Benefit Analysis
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration; Spinal Stenosis | interventions — Anesthesia, Epidural; Exercise; Ibuprofen; Cyclooxygenase 2 Inhibitors; aceclofenac; Anti-Inflammatory Agents, Non-Steroidal; Decompression; Gene Fusion; Codeine; Tramadol; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- HIVD-OP (Active Comparator): open or endoscopic discectomy
  Interventions: Procedure: open or endoscopic discectomy; Procedure: decompression; Procedure: instrumentation and fusion
- HIVD-NonOP (Experimental): epidural block, epidural adhesiolysis, exercise, ibuprofen, naxoprofen, Cox-2 inhibitor, aceclofenac, codeine, oxycontine, IRcodone, Tramadol
  Interventions: Procedure: epidural block; Other: exercise; Drug: ibuprofen, naxoprofen, Cox-2 inhibitor, aceclofenac; Drug: codeine, oxycontine, IRcodone, Tramadol; Procedure: epidural adhesiolysis
- LSS w/o instability -OP (Active Comparator): decompression, instrumentation and fusion
  Interventions: Procedure: decompression; Procedure: instrumentation and fusion
- LSS w/o instability -NonOP (Experimental): epidural block, epidural adhesiolysis, exercise, ibuprofen, naxoprofen, Cox-2 inhibitor, aceclofenac, codeine, oxycontine, IRcodone, Tramadol
  Interventions: Procedure: epidural block; Other: exercise; Drug: ibuprofen, naxoprofen, Cox-2 inhibitor, aceclofenac; Drug: codeine, oxycontine, IRcodone, Tramadol; Procedure: epidural adhesiolysis
- LSS w/ instability - OP (Active Comparator): decompression, instrumentation and fusion
  Interventions: Procedure: decompression; Procedure: instrumentation and fusion
- LSS w/ instability - NonOP (Experimental): epidural block, epidural adhesiolysis, exercise, ibuprofen, naxoprofen, Cox-2 inhibitor, aceclofenac, codeine, oxycontine, IRcodone, Tramadol
  Interventions: Procedure: epidural block; Other: exercise; Drug: ibuprofen, naxoprofen, Cox-2 inhibitor, aceclofenac; Drug: codeine, oxycontine, IRcodone, Tramadol; Procedure: epidural adhesiolysis
- No intervention group (Active Comparator): exercise, ibuprofen, naxoprofen, Cox-2 inhibitor, aceclofenac, codeine, oxycontine, IRcodone, Tramadol
  Interventions: Other: exercise; Drug: ibuprofen, naxoprofen, Cox-2 inhibitor, aceclofenac; Drug: codeine, oxycontine, IRcodone, Tramadol; Procedure: epidural adhesiolysis
- Intervention group (Experimental): epidural block, epidural adhesiolysis
  Interventions: Procedure: epidural block

INTERVENTIONS:
Procedure: open or endoscopic discectomy — FDA approved surgical procedures
  Arms: HIVD-OP
Procedure: epidural block — epidural block
  Arms: HIVD-NonOP; Intervention group; LSS w/ instability - NonOP; LSS w/o instability -NonOP
Other: exercise — educated exercise
  Arms: HIVD-NonOP; LSS w/ instability - NonOP; LSS w/o instability -NonOP; No intervention group
Drug: ibuprofen, naxoprofen, Cox-2 inhibitor, aceclofenac — FDA approved medication such as ibuprofen, naxoprofen etc.
  Other Names: NSAID
  Arms: HIVD-NonOP; LSS w/ instability - NonOP; LSS w/o instability -NonOP; No intervention group
Procedure: decompression — FDA approved surgical procedure such as lamiectom and, laminotomy
  Arms: HIVD-OP; LSS w/ instability - OP; LSS w/o instability -OP
Procedure: instrumentation and fusion — FDA approved surgical procedure such as PLIF, ALIF, DLIF, OLI and TLIF
  Arms: HIVD-OP; LSS w/ instability - OP; LSS w/o instability -OP
Drug: codeine, oxycontine, IRcodone, Tramadol — FDA approved opioid drug such as codeine, oxycontin, IRcodon
  Other Names: opioid
  Arms: HIVD-NonOP; LSS w/ instability - NonOP; LSS w/o instability -NonOP; No intervention group
Procedure: epidural adhesiolysis — FDA approved epidural adhesiolysis with catheter or endoscope
  Arms: HIVD-NonOP; LSS w/ instability - NonOP; LSS w/o instability -NonOP; No intervention group

SUMMARY:
Purpose: Comparative effectiveness research (CER) between surgical and non-surgical treatment for patients with low back pain Hypothesis: There will be significant differences in surgical and non-surgical treatment effect in patients who need operation for herniated intervertebral disc and spinal stenosis.

DETAILED DESCRIPTION:
Background: Eighty percents of the total population experiences lower back pain (LBP). Prevalence of LBP is about 20 to 30%. LBP is the most frequent disease and causes a lot of the medical and social costs. Recently the traditional drug therapy, exercise therapy has been developed and various non-surgical treatments have been developed. Surgical techniques are also rapidly evolving. In Korea lumbar spine surgeries were performed in accordance with the national practice guidelines presented by the Health Insurance Review and Assessment Service. Many patients who do not meet the surgical criteria undergo the non-surgical treatment, but there is no reliable research data for a systematic and cost-effective results of non-surgical treatment. It will be a big part of the future medical expenses because there is no guideline for the expensive procedure.

Contents:

1. Prospective randomized controlled trials to evaluate effectiveness and efficacy between surgical vs. non-surgical treatment for optimal treatment of low back pain
2. Prospective observational clinical study for non-surgical treatment methods
3. Analysis of health insurance data
4. Comprehensive symposium
5. Provide guideline for optimal treatment of low back pain
6. The results will be used to reflect National health insurance policy Development Results: Suggestion of guideline for optimal treatment of low back pain through analysis of efficacy and effectiveness between treatments

ELIGIBILITY:
Inclusion Criteria:

1. Herniated intervertebral disease, Low back pain over 6 weeks: if neurological deficit is combined early surgery is allowed; Over 18 years; Visual analogue pain score over 5; Compatible findings in MRI and/or CT
2. Lumbar spinal stenosis without instability, Low back pain over 3 months: if neurological deficit is combined early surgery is allowed; Over 18 years; Visual analogue pain score over 5; Compatible findings in MRI and/or CT; Without instability (15 degrees and 4mm motion)
3. Lumbar spinal stenosis with instability, Low back pain over 3 months: if neurological deficit is combined early surgery is allowed; Over 18 years; Visual analogue pain score over 5; Compatible findings in MRI and/or CT; With instability (15 degrees and 4mm motion)
4. No surgical indication, Low back pain over 6 weeks: if neurological deficit is combined early surgery is allowed; Over 18 years; Visual analogue pain score over 5; Compatible findings in MRI and/or CT;

Exclusion Criteria:

1. Herniated intervertebral disease, Cauda equine syndrome; Instability (15degrees, 4mm motion); Fracture, pregnancy; Any comorbidities that preclude operation; Combined disease: Neuromuscular disease, parkinson's disease, inflammatory arthritis, symptomatic spinal tumor, myelopathy, spinal infection; Previous lumbar spinal surgery; Neurological deficit that necessitates surgery
2. Lumbar spinal stenosis without instability, Cauda equine syndrome; Instability (15degrees, 4mm motion); Fracture, pregnancy Any comorbidities that preclude operation; Combined disease: Neuromuscular disease, parkinson's disease, inflammatory arthritis, symptomatic spinal tumor, myelopathy, spinal infection; Previous lumbar spinal surgery; Neurological deficit that necessitates surgery
3. Lumbar spinal stenosis with instability, Cauda equine syndrome; Fracture, pregnancy; Any comorbidities that preclude operation; Combined disease: Neuromuscular disease, parkinson's disease, inflammatory arthritis, symptomatic spinal tumor, myelopathy, spinal infection Previous lumbar spinal surgery; Neurological deficit that necessitates surgery
4. No surgical indication, Cauda equine syndrome; Fracture, pregnancy; Combined disease: Neuromuscular disease, parkinson's disease, inflammatory arthritis, symptomatic spinal tumor, myelopathy, spinal infection; Neurological deficit that necessitates surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1102 (Actual)
Dates: Start 2016-09; Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Compare the change of pain score after treatment | baseline and 24 months after treatment.
  Visual analog scale (VAS) is decresed more than 2.5 or VAS is less than 3.5.

SECONDARY OUTCOMES:
Appropriate conservative treatment period | 1, 3, 6, 12, 24 months after treatment.
  Appropriate conservative treatment period, Cost-effectiveness analysis (Quality of life index (SF-36, EQ-5D-5L), Direct medical cost)
the change of pain score (Visual anlogue pain score) after time of treatment | 1, 3, 6, 12, 24 months after treatment.
  compare the trend of change with mixed-model
Cost-effectiveness | 24 month after treatment
  Compare direct cost after each treatment
Quality of life index (SF-36) | 1, 3, 6, 12, 24 months after treatment.
  compare the trend of change with mixed-model
Quality of life index (EQ-5D-5L) | 1, 3, 6, 12, 24 months after treatment.
  compare the trend of change with mixed-model

CONTACTS AND LOCATIONS:
Overall Officials: Chun Kee Chung, Professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided